CLINICAL TRIAL: NCT05110131
Title: Comparison and Synergistic Evaluation of Needle Aspiration and Forceps Biopsy for Diagnosis of Lung Lesions With Electromagnetic Navigation Bronchoscopy
Brief Title: Evaluation of the Synergistic Impact of Needle and Forceps Biopsy With Electromagnetic Navigation Bronchoscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Yeon Wook Kim, Prof., Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CONFIDENT_ENB
Record Dates: First submitted 2021-10-14; First posted 2021-11-05 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Lung Cancer (Diagnosis)
Keywords: Electromagnetic Navigation Bronchoscopy; Bronchoscopy; Diagnosis
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Who Masked: Participant, Care Provider, Investigator
Masking Description: The attending physician and patient will be blinded to the randomized group and which method of biopsy (needle or forceps) would be performed first. The pulmonologist performing the ENB procedure will be informed just before the start of the procedure which group the patient is affiliated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needle-first (Active Comparator): Participants affiliated to this arm will undergo ENB-guided biopsy with needle aspiration first, followed by forceps biopsy
  Interventions: Device: Device for performing biopsy via electromagnetic navigation bronchoscopy
- Forceps-first (Active Comparator): Participants affiliated to this arm will undergo ENB-guided biopsy with forceps first, followed by needle aspiration.
  Interventions: Device: Device for performing biopsy via electromagnetic navigation bronchoscopy

INTERVENTIONS:
Device: Device for performing biopsy via electromagnetic navigation bronchoscopy — Device for performing biopsy via electromagnetic navigation bronchoscopy (needle and forceps)

SUMMARY:
This randomized crossover study aimed to evaluate whether a multimodal biopsy strategy using both needle and forceps can provide additive benefits compared with a single device for diagnosing peripheral pulmonary lesions with electromagnetic navigation bronchoscopy under moderate sedation and assess the comparative yield and discordance between the two devices.

DETAILED DESCRIPTION:
This randomized crossover study aimed to evaluate whether combining electromagnetic navigation bronchoscopy (ENB)-guided needle aspiration and forceps biopsy provides synergistic benefits, and compare the diagnostic performance of needle aspiration biopsy and forceps biopsy for diagnosis of pulmonary lesions.

The investigators designed this study to prospectively enroll patients with lung lesions that warrant histologic diagnosis and are feasible for undergoing electromagnetic bronchoscopy under moderate sedation. Participants will be randomized to two groups. One group will receive an ENB-guided biopsy with lung lesion with needle aspiration followed by forceps biopsy (needle-first group), while the other groups will receive the same procedure with forceps biopsy followed by needle aspiration biopsy (forceps-first group). All participants will undergo ENB under moderate sedation without the concurrent use of other guiding techniques such as fluoroscopy and radial endobronchial sonography. All participants will be followed up for up to 12 months to confirm the final diagnosis.

The primary endpoint is the diagnostic accuracy of combined needle aspiration and forceps biopsy for diagnosing pulmonary lesions compared with forceps biopsy alone. Diagnostic accuracy was defined as the proportion of participants in whom the biopsy yielded a definitive diagnosis, consistent with the strict definition; a biopsy procedure was considered diagnostic if the specimen established a definitive malignancy (true positive) or a specific benign diagnosis that sufficiently represented the lesion and informed further management (true negative) without the change in diagnosis through 12 months of follow-up.

Secondary endpoints include diagnostic accuracy of the combination compared with needle aspiration alone, sensitivity for malignancy, and the strictly defined diagnostic yield determined solely based on the ENB procedural encounter, successful lesion approach, sampling duration, number of attempts for needle and forceps biopsy, and adverse events related to the ENB procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung lesions with a possibility of malignancy and need tissue confirmation, which is eligible for ENB procedure under moderate sedation

Exclusion Criteria:

* Patients who disagree to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2024-11-13 (Estimated)

PRIMARY OUTCOMES:
Conservative diagnostic accuracy at 12 months | Confirmed by follow-up results at 12 months
  ([True positive + True negative]/All biopsied performed)

SECONDARY OUTCOMES:
Sensitivity of needle or forceps biopsy for diagnosis of malignancy | Confirmed by follow-up results at 12 months
  True positive/Confirmed malignancy cases
Diagnostic yield at index procedure | At index procedure
  The proportion of pathologic results that leads to a specific malignant or benign diagnosis
Duration of procedure | At index procedure
  Total duration and time per sampling for needle and forceps biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Yeon Wook Kim, MD., PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Folch EE, Pritchett MA, Nead MA, Bowling MR, Murgu SD, Krimsky WS, Murillo BA, LeMense GP, Minnich DJ, Bansal S, Ellis BQ, Mahajan AK, Gildea TR, Bechara RI, Sztejman E, Flandes J, Rickman OB, Benzaquen S, Hogarth DK, Linden PA, Wahidi MM, Mattingley JS, Hood KL, Lin H, Wolvers JJ, Khandhar SJ; NAVIGATE Study Investigators. Electromagnetic Navigation Bronchoscopy for Peripheral Pulmonary Lesions: One-Year Results of the Prospective, Multicenter NAVIGATE Study. J Thorac Oncol. 2019 Mar;14(3):445-458. doi: 10.1016/j.jtho.2018.11.013. Epub 2018 Nov 23. PMID 30476574
- [Background] Vachani A, Maldonado F, Laxmanan B, Kalsekar I, Murgu S. The Impact of Alternative Approaches to Diagnostic Yield Calculation in Studies of Bronchoscopy. Chest. 2022 May;161(5):1426-1428. doi: 10.1016/j.chest.2021.08.074. Epub 2021 Sep 7. No abstract available. PMID 34506792
- [Background] Ost DE, Ernst A, Lei X, Kovitz KL, Benzaquen S, Diaz-Mendoza J, Greenhill S, Toth J, Feller-Kopman D, Puchalski J, Baram D, Karunakara R, Jimenez CA, Filner JJ, Morice RC, Eapen GA, Michaud GC, Estrada-Y-Martin RM, Rafeq S, Grosu HB, Ray C, Gilbert CR, Yarmus LB, Simoff M; AQuIRE Bronchoscopy Registry. Diagnostic Yield and Complications of Bronchoscopy for Peripheral Lung Lesions. Results of the AQuIRE Registry. Am J Respir Crit Care Med. 2016 Jan 1;193(1):68-77. doi: 10.1164/rccm.201507-1332OC. PMID 26367186
- [Background] Gildea TR, Folch EE, Khandhar SJ, Pritchett MA, LeMense GP, Linden PA, Arenberg DA, Rickman OB, Mahajan AK, Singh J, Cicenia J, Mehta AC, Lin H, Mattingley JS; NAVIGATE Study Investigators. The Impact of Biopsy Tool Choice and Rapid On-Site Evaluation on Diagnostic Accuracy for Malignant Lesions in the Prospective: Multicenter NAVIGATE Study. J Bronchology Interv Pulmonol. 2021 Jul 1;28(3):174-183. doi: 10.1097/LBR.0000000000000740. PMID 33369988
- [Background] Folch EE, Labarca G, Ospina-Delgado D, Kheir F, Majid A, Khandhar SJ, Mehta HJ, Jantz MA, Fernandez-Bussy S. Sensitivity and Safety of Electromagnetic Navigation Bronchoscopy for Lung Cancer Diagnosis: Systematic Review and Meta-analysis. Chest. 2020 Oct;158(4):1753-1769. doi: 10.1016/j.chest.2020.05.534. Epub 2020 May 23. PMID 32450240
- [Background] Mondoni M, Sotgiu G, Bonifazi M, Dore S, Parazzini EM, Carlucci P, Gasparini S, Centanni S. Transbronchial needle aspiration in peripheral pulmonary lesions: a systematic review and meta-analysis. Eur Respir J. 2016 Jul;48(1):196-204. doi: 10.1183/13993003.00051-2016. Epub 2016 May 12. PMID 27174878
- [Derived] Kim YW, Kim HJ, Kwon BS, Lee YJ, Song MJ, Yoon SH, Lim SY, Lee YJ, Park JS, Cho YJ, Lee KH, Chung JH, Han YB, Maldonado F, Ahn SY, Park Y, Joo DH, Lee JH, Lee CT. Diagnostic Yield and Synergistic Impact of Needle Aspiration and Forceps Biopsy With Electromagnetic Navigation Bronchoscopy for Peripheral Pulmonary Lesions: A Randomized Controlled Trial. Chest. 2025 Jul;168(1):236-247. doi: 10.1016/j.chest.2025.02.015. Epub 2025 Feb 22. PMID 39993594
- [Derived] Kim YW, Kim HJ, Yoon SH, Lee KH, Park YM, Ahn SY, Song MJ, Kwon BS, Lim SY, Lee YJ, Park JS, Cho YJ, Yoon HI, Lee JH, Lee CT. Evaluation of the synergistic impact of needle and forceps biopsy with electromagnetic navigation bronchoscopy: the CONFIDENT-ENB trial design. BMC Pulm Med. 2022 Aug 19;22(1):319. doi: 10.1186/s12890-022-02104-w. PMID 35986257